CLINICAL TRIAL: NCT04856683
Title: PRecisiOn MEdicine to Target Frailty of Endocrine-metabolic Origin
Acronym: PROMETEO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Andrea M. Isidori, Full Professor, University of Roma La Sapienza
Other Study IDs: PROMETEO
Record Dates: First submitted 2021-04-13; First posted 2021-04-23 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Frailty
Keywords: Adrenal disorders; Gonadal disorders; Type 2 diabetes mellitus; Pituitary disorders; Bone disorders; Biostatistics/bioinformatics
MeSH Terms: conditions — Frailty; Adrenal Gland Diseases; Gonadal Disorders; Diabetes Mellitus, Type 2; Pituitary Diseases; Bone Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with endocrine and metabolic diseases: Patients with endocrine and metabolic diseases (hypothalamic-pituitary-gonadal and adrenal diseases, type 2 diabetes mellitus and bone diseases)

SUMMARY:
This is a multicenter, observational, retrospective and prospective study for the evaluation of precision medicine to target frailty of endocrine-metabolic origin, with a genetic study.

DETAILED DESCRIPTION:
Overall summary Frailty results from the lifelong accumulation of damage caused by age- and disease-related impairment of the repair network. The amount of cellular damage needed to alter function is uncertain and determined on an individual basis. Assessing cumulative dysfunction in different systems (hormonal, metabolic, immune, cardiovascular, and skeletal) is crucial as the relationship with frailty is nonlinear and not linked to the severity in one system. When subtle, declining functions reaches an aggregate crucial level, and frailty becomes evident. The frail individual is who, after a mild stressor event, undergoes a larger deterioration, which manifest as functional dependency (hospitalization), and who does not return to baseline homoeostasis (favoring polypharmacy). By implementing precision medicine, retrospective and prospective data collected in five referral centers covering densely populated regions in Italy, will be merged and thoroughly analyzed. This network aims at identifying novel biomarkers, predictors of treatment response, and simplified management for complex multiple endocrine comorbidities. The network will investigate emerging and highly prevalent disorders linked to frailty: the gonadal and adrenal, metabolic, neuroendocrine, skeletal. The network will generate scores and precision-medicine based algorithms for the fragile population, often excluded from clinical trials while absorbing most of healthcare expenditure.

Background Frailty is raising globally. Patients with multiple endocrine and metabolic comorbidities (MEDs) are at high risk for inappropriate prescriptions, with negative effects on health outcomes and costs. Endocrine and metabolic comorbidities often coexist with frailty being the common endpoint in patients requiring intensive medical care (falls, disability, hospitalization, and mortality). Concomitant multiple medications aggravate frailty by increasing the risk of interactions, adverse effects and reduce efficacy. The cost of supporting these high-risk population are no longer sustainable for the National Health System (NHS). The pathophysiology of frailty is poorly understood, but multiple endocrine dysfunctions are often associated. Dysregulation of the hypothalamic-pituitary-gonadal and adrenal axes are often associated with metabolic disease (Type 2 Diabetes Mellitus-T2D) as well as bone diseases. In 2018 data from the European Male Aging Study (EMAS) showed that both androgen and nonandrogenic anabolic hormones were independently associated with change in frailty status. Other studies showed that frailty was independently associated with chronically raised diurnal cortisol. Diabetes and osteoporosis (OP) are commonly associated with a significant health burden, especially in elderly individuals. Diabetes is also associated with a wide spectrum of comorbidities (cardiovascular disease, impairment of bone quality, hypogonadism, reduced quality of life, obesity). OP is a complex disorder whose pathogenesis is due to the interaction of various predisposing genetic and epigenetic factors regulating bone and mineral metabolism and non-skeletal risk factors that could influence the risk of fall. Genome-wide association studies (GWAS), epigenetic factors and circulating micro-RNA have opened new horizons for the discovery of genetic loci and variants associated with OP and fracture risk, identifying replicated genetic loci associated with OP. Circulating microRNA profiles have also a prognostic value making them attractive, blood-based, non-invasive biomarkers for prediction and staging of endocrine diseases. Moreover, evidence suggests that inflammation has a major role in the pathophysiology of frailty through an abnormal, low-grade inflammatory chronic response that is hyper-responsive to stimuli. Several inflammatory cytokines have been independently associated with frailty and a link was demonstrated between immune cell function and steroid hormone levels in the recently published DREAM trial. Response to therapy in T2D is often patient-related especially in frail patients. However specific biomarkers are needed for disease monitoring and prediction of disease progression or therapy response. Finally, pituitary diseases are associated with increased mortality and morbidity. This can be a direct effect of hormonal hypersecretion but also secondary to hypopituitarism (HP) caused by mass effect, or a direct consequence of trauma, as well as an important side effect of the treatment itself on pituitary lesions (novel immune check-point inhibitors). HP is globally under-diagnosed and insidious with tremendous effects on quality of life (QoL) as well. All the above mentioned and several other studies suggest an important role of the endocrine system on the development of frailty. It is very likely that comorbidities and drugs can accelerate the frailty of endocrine and metabolic origin. Finally, as concern inappropriate prescriptions, some algorithms were demonstrated particularly reliable. Combining clinical, epidemiological, social, hospital admissions and drug prescription data, has been proven a valid approach to identify inappropriate prescriptions due to drug ineffectiveness and to evaluate cost of polypharmacy.

Hypothesis and Significance Dysregulation of glucocorticoid secretion and hypogonadism due to primary adrenal or gonadal disorders are independent contributors to frailty and failure to treat effectively cardiovascular, metabolic and bone diseases. Prompt restoration of gonadal and adrenal function, when altered, can reduce the need for multi-drug prescription necessary to target high blood pressure, cardiovascular remodeling, osteoporosis and diabetes mellitus.

Less than 50% of patients with T2D had good glycemic control, understanding the mechanisms of Dipeptidyl peptidase-4 (DPP4) inhibitors and Glucagon-like peptide 1 (GLP1)-receptor agonist therapy is needed to predict the response to treatment. Genetic analysis and circulating microRNA profiling may help choosing the appropriate glucose-lowering drugs in T2D patients.

The high prevalence of pituitary and neuroendocrine disorders has a significant impact on morbidity, mortality and QoL. Tailoring diagnostic and therapeutic strategies will lead to early diagnosis of these diseases and their complications allowing to select the best long-term management.

A correlation between genetic and epigenetic risk of OP and fragility fractures (FF), two major components of frailty, is hypothesized and the investigators aim to identify early the subjects at higher risk and predict their response to anti-fracture drug.

Some complex endocrine disorders require extensive use of healthcare resources. Health Care Utilization (HCU) data offer accurate information on the prevalence, incidence, and duration of drugs use providing a comprehensive picture of the therapeutic habits. Linking prescription and clinical-administrative data could allow this network to investigate the inappropriate prescription patterns and the association with worse clinical outcomes.

Implications of the Study The case load of hospital care, diagnostic procedures and drug costs for non-communicable diseases is exceeding sustainability in all countries with a negative impact on public health system. The exponential rise in costs is due to the ageing of the population, prevalence of chronic disorders, improved acute care and new expensive drugs. Rationalization of expenditures is mandatory. Personalize diagnostic procedures, therapeutic approaches and management of comorbidities in highly prevalent disorders is only the immediately sustainable approach. The endocrine and metabolic disorders offer the ideal model to quantify the advantages of shifting from a non-personalized approached to precision etiological treatment strategies. This can lead to a rapid and substantial decline in cost expenditure in terms of number of hospital access, prescribed investigations, and inappropriate medication use. Expected outcomes is a reduction of NIH cost due to saving in 1) polypharmacy and 2) reduced hospitalization for the greater efficacy of drugs prescribed using and personalized algorithm, 3) reduced side effects due to multiple-drug interactions.

ELIGIBILITY:
Inclusion Criteria:

* presence of endocrine and metabolic diseases (hypothalamic-pituitary-gonadal and adrenal diseases, type 2 diabetes mellitus, and bone diseases);
* signed informed consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with endocrine and metabolic diseases (hypothalamic-pituitary-gonadal and adrenal diseases, type 2 diabetes mellitus and bone diseases).
  Retrospective cohort of 1100 subjects randomly selected from the 2000 on-file, after matching inclusion criteria.
  Prospective cohort of 378 subjects from the 1100 patients recruited in the retrospective phase.
Sampling Method: Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2020-08-10 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2024-08-09 (Estimated)

PRIMARY OUTCOMES:
Composite Clinical Score | Baseline
  To derive a Composite Clinical Score able to identify endocrine fragile patients (occurrence of at least one of the following events: falls, disability, hospitalization, and mortality within the previous 18-months).
Prediction of frailty | Baseline
  Validation of Composite Clinical Score to predict frailty occurrence

SECONDARY OUTCOMES:
Peripheral blood mononuclear cell subpopulations | Baseline
  Number of cells (number per mm3) of peripheral blood mononuclear cell subpopulations
Molecular profiling | Baseline
  Circulating miRNA in blood samples from patients with adrenal and gonadal diseases
Steroid profiling | Baseline
  Steroid metabolites assessed by liquid chromatography-mass spectrometry (LC-MS/MS)
Measure of vascular flows though contrast enhanced ultrasound in endocrine glands | Baseline
  Coupling vascular glandular inflow with hormonal outflow
Measure of liver vascular inflow through 4 dimensional (4D)-flow MRI | Baseline
  Coupling liver vascular inflow with liver glucocorticoid metabolism
Serotonin Transporter 5-HTTLPR polymorphism | Baseline
  To study the effects of Serotonin Transporter 5-HTTLPR polymorphism on gastrointestinal intolerance to metformin in a population of T2D subjects and its relationship with glycometabolic control
Circulating microRNAs | Baseline and post 6 months
  To evaluate circulating microRNAs in blood samples from patients with T2D before and after GLP1-receptor agonist or DPP4 inhibitors therapy, in order to identify markers predicting treatment response, therapeutic efficacy and side effects
Gene polymorphisms | Baseline and post 6 months
  To evaluate gene polymorphisms in blood samples from patients with T2D before and after GLP1-RA or DPP4 inhibitors therapy, in order to identify markers predicting treatment response, therapeutic efficacy and side effects
Cardio-metabolic stratification risk | Baseline
  To elaborate a risk stratification approach for cardiovascular, metabolic and cerebrovascular outcomes in pituitary patients aimed to personalize treatment and follow-up in pituitary diseases.
Psychological function | Baseline
  Psychological function assessed by QoL questionnaire in pituitary diseases
Osteoporosis stratification risk | Baseline
  Gene analysis to elaborate a risk screening panel for osteoporosis
Epigenetic biomarkers | Baseline
  To individuate possible serum epigenetic biomarkers of osteoporosis status and fragility fractures risk
Multiple endocrine and metabolic comorbidities | Baseline
  To identify patients with multiple endocrine and metabolic comorbidities and assess the incidence of major clinical events using regional registries
Inappropriate therapeutic regimen | Baseline
  To individuate inappropriate therapeutic regimen (drug prescriptions or suboptimal adherence) in patients with multiple endocrine and metabolic comorbidities

CONTACTS AND LOCATIONS:
Overall Officials: Andrea M Isidori, Prof, Principal Investigator — Department of Experimental Medicine, "Sapienza" University of Rome
Locations (5):
- Italy (5):
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliero-Universitaria Policlinico Umberto I, Rome
  - Ospedale San Giovanni Calibita-Fatebenefratelli Fondazione Fatebenefratelli per la Ricerca e la Formazione Sanitaria e Sociale, Rome
  - Azienda Ospedaliero-Universitaria Senese, Siena

REFERENCES:
- [Background] Finkelstein J, Friedman C, Hripcsak G, Cabrera M. Potential utility of precision medicine for older adults with polypharmacy: a case series study. Pharmgenomics Pers Med. 2016 Apr 15;9:31-45. doi: 10.2147/PGPM.S101474. eCollection 2016. PMID 27143951
- [Background] Joseph SM, Rich MW. Targeting Frailty in Heart Failure. Curr Treat Options Cardiovasc Med. 2017 Apr;19(4):31. doi: 10.1007/s11936-017-0527-5. PMID 28357683
- [Background] Morley JE. Hormones and Sarcopenia. Curr Pharm Des. 2017 Nov 28;23(30):4484-4492. doi: 10.2174/1381612823666161123150032. PMID 27881060
- [Background] Swiecicka A, Eendebak RJAH, Lunt M, O'Neill TW, Bartfai G, Casanueva FF, Forti G, Giwercman A, Han TS, Slowikowska-Hilczer J, Lean MEJ, Pendleton N, Punab M, Vanderschueren D, Huhtaniemi IT, Wu FCW, Rutter MK; European Male Ageing Study Group. Reproductive Hormone Levels Predict Changes in Frailty Status in Community-Dwelling Older Men: European Male Ageing Study Prospective Data. J Clin Endocrinol Metab. 2018 Feb 1;103(2):701-709. doi: 10.1210/jc.2017-01172. PMID 29186457
- [Background] Saad F, Rohrig G, von Haehling S, Traish A. Testosterone Deficiency and Testosterone Treatment in Older Men. Gerontology. 2017;63(2):144-156. doi: 10.1159/000452499. Epub 2016 Nov 18. PMID 27855417
- [Background] Ladapo JA, Budoff MJ, Sharp D, Kuo JZ, Huang L, Maniet B, Herman L, Monane M. Utility of a Precision Medicine Test in Elderly Adults with Symptoms Suggestive of Coronary Artery Disease. J Am Geriatr Soc. 2018 Feb;66(2):309-315. doi: 10.1111/jgs.15215. Epub 2017 Dec 6. PMID 29210056
- [Background] Ramaswami R, Bayer R, Galea S. Precision Medicine from a Public Health Perspective. Annu Rev Public Health. 2018 Apr 1;39:153-168. doi: 10.1146/annurev-publhealth-040617-014158. Epub 2017 Nov 20. PMID 29166244
- [Background] Kane AE, Gregson E, Theou O, Rockwood K, Howlett SE. The association between frailty, the metabolic syndrome, and mortality over the lifespan. Geroscience. 2017 Apr;39(2):221-229. doi: 10.1007/s11357-017-9967-9. Epub 2017 Mar 9. PMID 28281219
- [Background] Johar H, Emeny RT, Bidlingmaier M, Reincke M, Thorand B, Peters A, Heier M, Ladwig KH. Blunted diurnal cortisol pattern is associated with frailty: a cross-sectional study of 745 participants aged 65 to 90 years. J Clin Endocrinol Metab. 2014 Mar;99(3):E464-8. doi: 10.1210/jc.2013-3079. Epub 2014 Feb 24. PMID 24564322
- [Background] Clegg A, Young J, Iliffe S, Rikkert MO, Rockwood K. Frailty in elderly people. Lancet. 2013 Mar 2;381(9868):752-62. doi: 10.1016/S0140-6736(12)62167-9. Epub 2013 Feb 8. PMID 23395245
- [Background] Isidori AM, Venneri MA, Graziadio C, Simeoli C, Fiore D, Hasenmajer V, Sbardella E, Gianfrilli D, Pozza C, Pasqualetti P, Morrone S, Santoni A, Naro F, Colao A, Pivonello R, Lenzi A. Effect of once-daily, modified-release hydrocortisone versus standard glucocorticoid therapy on metabolism and innate immunity in patients with adrenal insufficiency (DREAM): a single-blind, randomised controlled trial. Lancet Diabetes Endocrinol. 2018 Mar;6(3):173-185. doi: 10.1016/S2213-8587(17)30398-4. Epub 2017 Dec 8. PMID 29229498
- [Background] DeFronzo RA. Pathogenesis of type 2 diabetes mellitus. Med Clin North Am. 2004 Jul;88(4):787-835, ix. doi: 10.1016/j.mcna.2004.04.013. PMID 15308380
- [Background] Intensive blood-glucose control with sulphonylureas or insulin compared with conventional treatment and risk of complications in patients with type 2 diabetes (UKPDS 33). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):837-53. PMID 9742976
- [Background] Rossi MC, Nicolucci A, Arcangeli A, Cimino A, De Bigontina G, Giorda C, Meloncelli I, Pellegrini F, Valentini U, Vespasiani G; Associazione Medici Diabetologi Annals Study Group. Baseline quality-of-care data from a quality-improvement program implemented by a network of diabetes outpatient clinics. Diabetes Care. 2008 Nov;31(11):2166-8. doi: 10.2337/dc08-0469. Epub 2008 Aug 11. PMID 18694979
- [Background] Dujic T, Zhou K, Tavendale R, Palmer CN, Pearson ER. Effect of Serotonin Transporter 5-HTTLPR Polymorphism on Gastrointestinal Intolerance to Metformin: A GoDARTS Study. Diabetes Care. 2016 Nov;39(11):1896-1901. doi: 10.2337/dc16-0706. Epub 2016 Aug 4. PMID 27493135
- [Background] Guay C, Regazzi R. Circulating microRNAs as novel biomarkers for diabetes mellitus. Nat Rev Endocrinol. 2013 Sep;9(9):513-21. doi: 10.1038/nrendo.2013.86. Epub 2013 Apr 30. PMID 23629540
- [Background] Sebastiani G, Nigi L, Grieco GE, Mancarella F, Ventriglia G, Dotta F. Circulating microRNAs and diabetes mellitus: a novel tool for disease prediction, diagnosis, and staging? J Endocrinol Invest. 2017 Jun;40(6):591-610. doi: 10.1007/s40618-017-0611-4. Epub 2017 Feb 17. PMID 28213644
- [Background] Jamaluddin JL, Huri HZ, Vethakkan SR. Clinical and genetic predictors of dipeptidyl peptidase-4 inhibitor treatment response in Type 2 diabetes mellitus. Pharmacogenomics. 2016 Jun;17(8):867-81. doi: 10.2217/pgs-2016-0010. Epub 2016 Jun 1. PMID 27249660
- [Background] Catanzaro G, Besharat ZM, Chiacchiarini M, Abballe L, Sabato C, Vacca A, Borgiani P, Dotta F, Tesauro M, Po A, Ferretti E. Circulating MicroRNAs in Elderly Type 2 Diabetic Patients. Int J Endocrinol. 2018 Apr 10;2018:6872635. doi: 10.1155/2018/6872635. eCollection 2018. PMID 29849622
- [Background] Sherlock M, Ayuk J, Tomlinson JW, Toogood AA, Aragon-Alonso A, Sheppard MC, Bates AS, Stewart PM. Mortality in patients with pituitary disease. Endocr Rev. 2010 Jun;31(3):301-42. doi: 10.1210/er.2009-0033. Epub 2010 Jan 19. PMID 20086217
- [Background] Tanriverdi F, Schneider HJ, Aimaretti G, Masel BE, Casanueva FF, Kelestimur F. Pituitary dysfunction after traumatic brain injury: a clinical and pathophysiological approach. Endocr Rev. 2015 Jun;36(3):305-42. doi: 10.1210/er.2014-1065. Epub 2015 May 7. PMID 25950715
- [Background] Corsello SM, Barnabei A, Marchetti P, De Vecchis L, Salvatori R, Torino F. Endocrine side effects induced by immune checkpoint inhibitors. J Clin Endocrinol Metab. 2013 Apr;98(4):1361-75. doi: 10.1210/jc.2012-4075. Epub 2013 Mar 7. PMID 23471977
- [Background] Arosio M, Reimondo G, Malchiodi E, Berchialla P, Borraccino A, De Marinis L, Pivonello R, Grottoli S, Losa M, Cannavo S, Minuto F, Montini M, Bondanelli M, De Menis E, Martini C, Angeletti G, Velardo A, Peri A, Faustini-Fustini M, Tita P, Pigliaru F, Borretta G, Scaroni C, Bazzoni N, Bianchi A, Appetecchia M, Cavagnini F, Lombardi G, Ghigo E, Beck-Peccoz P, Colao A, Terzolo M; Italian Study Group of Acromegaly. Predictors of morbidity and mortality in acromegaly: an Italian survey. Eur J Endocrinol. 2012 Aug;167(2):189-98. doi: 10.1530/EJE-12-0084. Epub 2012 May 17. PMID 22596288
- [Background] Colao A, Ferone D, Marzullo P, Lombardi G. Systemic complications of acromegaly: epidemiology, pathogenesis, and management. Endocr Rev. 2004 Feb;25(1):102-52. doi: 10.1210/er.2002-0022. PMID 14769829
- [Background] Graversen D, Vestergaard P, Stochholm K, Gravholt CH, Jorgensen JO. Mortality in Cushing's syndrome: a systematic review and meta-analysis. Eur J Intern Med. 2012 Apr;23(3):278-82. doi: 10.1016/j.ejim.2011.10.013. Epub 2011 Nov 15. PMID 22385888
- [Background] Clayton RN, Raskauskiene D, Reulen RC, Jones PW. Mortality and morbidity in Cushing's disease over 50 years in Stoke-on-Trent, UK: audit and meta-analysis of literature. J Clin Endocrinol Metab. 2011 Mar;96(3):632-42. doi: 10.1210/jc.2010-1942. Epub 2010 Dec 30. PMID 21193542
- [Background] Mancini T, Kola B, Mantero F, Boscaro M, Arnaldi G. High cardiovascular risk in patients with Cushing's syndrome according to 1999 WHO/ISH guidelines. Clin Endocrinol (Oxf). 2004 Dec;61(6):768-77. doi: 10.1111/j.1365-2265.2004.02168.x. PMID 15579193
- [Background] Tomlinson JW, Holden N, Hills RK, Wheatley K, Clayton RN, Bates AS, Sheppard MC, Stewart PM. Association between premature mortality and hypopituitarism. West Midlands Prospective Hypopituitary Study Group. Lancet. 2001 Feb 10;357(9254):425-31. doi: 10.1016/s0140-6736(00)04006-x. PMID 11273062
- [Background] Mazziotti G, Chiavistelli S, Giustina A. Pituitary diseases and bone. Endocrinol Metab Clin North Am. 2015 Mar;44(1):171-80. doi: 10.1016/j.ecl.2014.10.014. Epub 2014 Nov 4. PMID 25732653
- [Background] Mazziotti G, Doga M, Frara S, Maffezzoni F, Porcelli T, Cerri L, Maroldi R, Giustina A. Incidence of morphometric vertebral fractures in adult patients with growth hormone deficiency. Endocrine. 2016 Apr;52(1):103-10. doi: 10.1007/s12020-015-0738-z. Epub 2015 Oct 3. PMID 26433736
- [Background] Mazziotti G, Frara S, Giustina A. Pituitary Diseases and Bone. Endocr Rev. 2018 Aug 1;39(4):440-488. doi: 10.1210/er.2018-00005. PMID 29684108
- [Background] Johnson MD, Woodburn CJ, Vance ML. Quality of life in patients with a pituitary adenoma. Pituitary. 2003 Sep;6(2):81-7. doi: 10.1023/b:pitu.0000004798.27230.ed. PMID 14703017
- [Background] Webb SM, Crespo I, Santos A, Resmini E, Aulinas A, Valassi E. MANAGEMENT OF ENDOCRINE DISEASE: Quality of life tools for the management of pituitary disease. Eur J Endocrinol. 2017 Jul;177(1):R13-R26. doi: 10.1530/EJE-17-0041. Epub 2017 Mar 28. PMID 28351913
- [Background] Andela CD, Scharloo M, Ramondt S, Tiemensma J, Husson O, Llahana S, Pereira AM, Kaptein AA, Kamminga NG, Biermasz NR. The development and validation of the Leiden Bother and Needs Questionnaire for patients with pituitary disease: the LBNQ-Pituitary. Pituitary. 2016 Jun;19(3):293-302. doi: 10.1007/s11102-016-0707-4. PMID 26809957
- [Background] Sonino N, Fava GA. Psychiatric disorders associated with Cushing's syndrome. Epidemiology, pathophysiology and treatment. CNS Drugs. 2001;15(5):361-73. doi: 10.2165/00023210-200115050-00003. PMID 11475942
- [Background] van Aken MO, Pereira AM, Biermasz NR, van Thiel SW, Hoftijzer HC, Smit JW, Roelfsema F, Lamberts SW, Romijn JA. Quality of life in patients after long-term biochemical cure of Cushing's disease. J Clin Endocrinol Metab. 2005 Jun;90(6):3279-86. doi: 10.1210/jc.2004-1375. Epub 2005 Mar 1. PMID 15741267
- [Background] Carosi G, Malchiodi E, Ferrante E, Sala E, Verrua E, Profka E, Giavoli C, Filopanti M, Beck-Peccoz P, Spada A, Mantovani G. Hypothalamic-Pituitary Axis in Non-Functioning Pituitary Adenomas: Focus on the Prevalence of Isolated Central Hypoadrenalism. Neuroendocrinology. 2015;102(4):267-273. doi: 10.1159/000430815. Epub 2015 Apr 29. PMID 25924873
- [Background] Terzolo M, Reimondo G, Berchialla P, Ferrante E, Malchiodi E, De Marinis L, Pivonello R, Grottoli S, Losa M, Cannavo S, Ferone D, Montini M, Bondanelli M, De Menis E, Martini C, Puxeddu E, Velardo A, Peri A, Faustini-Fustini M, Tita P, Pigliaru F, Peraga G, Borretta G, Scaroni C, Bazzoni N, Bianchi A, Berton A, Serban AL, Baldelli R, Fatti LM, Colao A, Arosio M; Italian Study Group of Acromegaly. Acromegaly is associated with increased cancer risk: a survey in Italy. Endocr Relat Cancer. 2017 Sep;24(9):495-504. doi: 10.1530/ERC-16-0553. Epub 2017 Jul 14. PMID 28710115
- [Background] Ronchi CL, Giavoli C, Ferrante E, Verrua E, Bergamaschi S, Ferrari DI, Corbetta S, Montefusco L, Arosio M, Ambrosi B, Spada A, Beck-Peccoz P. Prevalence of GH deficiency in cured acromegalic patients: impact of different previous treatments. Eur J Endocrinol. 2009 Jul;161(1):37-42. doi: 10.1530/EJE-09-0222. Epub 2009 Apr 7. PMID 19351744
- [Background] Giavoli C, Profka E, Verrua E, Ronchi CL, Ferrante E, Bergamaschi S, Sala E, Malchiodi E, Lania AG, Arosio M, Ambrosi B, Spada A, Beck-Peccoz P. GH replacement improves quality of life and metabolic parameters in cured acromegalic patients with growth hormone deficiency. J Clin Endocrinol Metab. 2012 Nov;97(11):3983-8. doi: 10.1210/jc.2012-2477. Epub 2012 Aug 17. PMID 22904173
- [Background] Chiodini I, Mascia ML, Muscarella S, Battista C, Minisola S, Arosio M, Santini SA, Guglielmi G, Carnevale V, Scillitani A. Subclinical hypercortisolism among outpatients referred for osteoporosis. Ann Intern Med. 2007 Oct 16;147(8):541-8. doi: 10.7326/0003-4819-147-8-200710160-00006. PMID 17938392
- [Background] Chiodini I, Torlontano M, Scillitani A, Arosio M, Bacci S, Di Lembo S, Epaminonda P, Augello G, Enrini R, Ambrosi B, Adda G, Trischitta V. Association of subclinical hypercortisolism with type 2 diabetes mellitus: a case-control study in hospitalized patients. Eur J Endocrinol. 2005 Dec;153(6):837-44. doi: 10.1530/eje.1.02045. PMID 16322389
- [Background] Chiodini I, Adda G, Scillitani A, Coletti F, Morelli V, Di Lembo S, Epaminonda P, Masserini B, Beck-Peccoz P, Orsi E, Ambrosi B, Arosio M. Cortisol secretion in patients with type 2 diabetes: relationship with chronic complications. Diabetes Care. 2007 Jan;30(1):83-8. doi: 10.2337/dc06-1267. PMID 17192338
- [Background] Zhukouskaya VV, Eller-Vainicher C, Gaudio A, Cairoli E, Ulivieri FM, Palmieri S, Morelli V, Orsi E, Masserini B, Barbieri AM, Polledri E, Fustinoni S, Spada A, Fiore CE, Chiodini I. In postmenopausal female subjects with type 2 diabetes mellitus, vertebral fractures are independently associated with cortisol secretion and sensitivity. J Clin Endocrinol Metab. 2015 Apr;100(4):1417-25. doi: 10.1210/jc.2014-4177. Epub 2015 Jan 15. PMID 25590217
- [Background] Ralston SH. Genetic determinants of susceptibility to osteoporosis. Curr Opin Pharmacol. 2003 Jun;3(3):286-90. doi: 10.1016/s1471-4892(03)00033-x. PMID 12810194
- [Background] Richards JB, Zheng HF, Spector TD. Genetics of osteoporosis from genome-wide association studies: advances and challenges. Nat Rev Genet. 2012 Jul 18;13(8):576-88. doi: 10.1038/nrg3228. PMID 22805710
- [Background] Arden NK, Baker J, Hogg C, Baan K, Spector TD. The heritability of bone mineral density, ultrasound of the calcaneus and hip axis length: a study of postmenopausal twins. J Bone Miner Res. 1996 Apr;11(4):530-4. doi: 10.1002/jbmr.5650110414. PMID 8992884
- [Background] Eisman JA. Genetics of osteoporosis. Endocr Rev. 1999 Dec;20(6):788-804. doi: 10.1210/edrv.20.6.0384. PMID 10605626
- [Background] Andrew T, Antioniades L, Scurrah KJ, Macgregor AJ, Spector TD. Risk of wrist fracture in women is heritable and is influenced by genes that are largely independent of those influencing BMD. J Bone Miner Res. 2005 Jan;20(1):67-74. doi: 10.1359/JBMR.041015. Epub 2004 Oct 25. PMID 15619671
- [Background] Rocha-Braz MG, Ferraz-de-Souza B. Genetics of osteoporosis: searching for candidate genes for bone fragility. Arch Endocrinol Metab. 2016 Aug;60(4):391-401. doi: 10.1590/2359-3997000000178. PMID 27533615
- [Background] Ioannidis JP, Ralston SH, Bennett ST, Brandi ML, Grinberg D, Karassa FB, Langdahl B, van Meurs JB, Mosekilde L, Scollen S, Albagha OM, Bustamante M, Carey AH, Dunning AM, Enjuanes A, van Leeuwen JP, Mavilia C, Masi L, McGuigan FE, Nogues X, Pols HA, Reid DM, Schuit SC, Sherlock RE, Uitterlinden AG; GENOMOS Study. Differential genetic effects of ESR1 gene polymorphisms on osteoporosis outcomes. JAMA. 2004 Nov 3;292(17):2105-14. doi: 10.1001/jama.292.17.2105. PMID 15523071
- [Background] Ralston SH, Uitterlinden AG, Brandi ML, Balcells S, Langdahl BL, Lips P, Lorenc R, Obermayer-Pietsch B, Scollen S, Bustamante M, Husted LB, Carey AH, Diez-Perez A, Dunning AM, Falchetti A, Karczmarewicz E, Kruk M, van Leeuwen JP, van Meurs JB, Mangion J, McGuigan FE, Mellibovsky L, del Monte F, Pols HA, Reeve J, Reid DM, Renner W, Rivadeneira F, van Schoor NM, Sherlock RE, Ioannidis JP; GENOMOS Investigators. Large-scale evidence for the effect of the COLIA1 Sp1 polymorphism on osteoporosis outcomes: the GENOMOS study. PLoS Med. 2006 Apr;3(4):e90. doi: 10.1371/journal.pmed.0030090. Epub 2006 Feb 21. PMID 16475872
- [Background] Uitterlinden AG, Ralston SH, Brandi ML, Carey AH, Grinberg D, Langdahl BL, Lips P, Lorenc R, Obermayer-Pietsch B, Reeve J, Reid DM, Amedei A, Bassiti A, Bustamante M, Husted LB, Diez-Perez A, Dobnig H, Dunning AM, Enjuanes A, Fahrleitner-Pammer A, Fang Y, Karczmarewicz E, Kruk M, van Leeuwen JP, Mavilia C, van Meurs JB, Mangion J, McGuigan FE, Pols HA, Renner W, Rivadeneira F, van Schoor NM, Scollen S, Sherlock RE, Ioannidis JP; APOSS Investigators; EPOS Investigators; EPOLOS Investigators; FAMOS Investigators; LASA Investigators; Rotterdam Study Investigators; GENOMOS Study. The association between common vitamin D receptor gene variations and osteoporosis: a participant-level meta-analysis. Ann Intern Med. 2006 Aug 15;145(4):255-64. doi: 10.7326/0003-4819-145-4-200608150-00005. PMID 16908916
- [Background] Langdahl BL, Uitterlinden AG, Ralston SH, Trikalinos TA, Balcells S, Brandi ML, Scollen S, Lips P, Lorenc R, Obermayer-Pietsch B, Reid DM, Armas JB, Arp PP, Bassiti A, Bustamante M, Husted LB, Carey AH, Perez Cano R, Dobnig H, Dunning AM, Fahrleitner-Pammer A, Falchetti A, Karczmarewicz E, Kruk M, van Leeuwen JP, Masi L, van Meurs JB, Mangion J, McGuigan FE, Mellibovsky L, Mosekilde L, Nogues X, Pols HA, Reeve J, Renner W, Rivadeneira F, van Schoor NM, Ioannidis JP; APOSS investigators; DOPS investigators; EPOS investigators; EPOLOS investigators; FAMOS investigators; LASA investigators; ERGO investigators; GENOMOS Study. Large-scale analysis of association between polymorphisms in the transforming growth factor beta 1 gene (TGFB1) and osteoporosis: the GENOMOS study. Bone. 2008 May;42(5):969-81. doi: 10.1016/j.bone.2007.11.007. Epub 2007 Dec 3. PMID 18284942
- [Background] van Meurs JB, Trikalinos TA, Ralston SH, Balcells S, Brandi ML, Brixen K, Kiel DP, Langdahl BL, Lips P, Ljunggren O, Lorenc R, Obermayer-Pietsch B, Ohlsson C, Pettersson U, Reid DM, Rousseau F, Scollen S, Van Hul W, Agueda L, Akesson K, Benevolenskaya LI, Ferrari SL, Hallmans G, Hofman A, Husted LB, Kruk M, Kaptoge S, Karasik D, Karlsson MK, Lorentzon M, Masi L, McGuigan FE, Mellstrom D, Mosekilde L, Nogues X, Pols HA, Reeve J, Renner W, Rivadeneira F, van Schoor NM, Weber K, Ioannidis JP, Uitterlinden AG; GENOMOS Study. Large-scale analysis of association between LRP5 and LRP6 variants and osteoporosis. JAMA. 2008 Mar 19;299(11):1277-90. doi: 10.1001/jama.299.11.1277. PMID 18349089